CLINICAL TRIAL: NCT01068392
Title: A Phase II Study of Oxaliplatin and Prednisolone (Ox-P) for Patients With Relapsed or Refractory Marginal Zone B-cell Lymphoma
Brief Title: Oxaliplatin and Prednisolone (Ox-P) for Patients With Relapsed or Refractory Marginal Zone B-cell Lymphoma(MZL)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dong-A University Hospital (Other)
Collaborators: Samsung Medical Center (Other); Asan Medical Center (Other); Chung-Ang University (Other); Kyungpook National University Hospital (Other); Chonnam National University Hospital (Other); Korea Cancer Center Hospital (Other); Korea University (Other)
Responsible Party: Principal Investigator, Sung Yong Oh, Department of internal medicine, Dong-A University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CISL-MZL-10-3
Record Dates: First submitted 2010-02-11; First posted 2010-02-12 (Estimated); Last update posted 2014-11-04 (Estimated); Status verified 2014-11

CONDITIONS: B-cell Lymphomas
Keywords: relapsed; marginal zone B-cell lymphoma; oxaliplatin; prednisolone
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence; Lymphoma, B-Cell, Marginal Zone | interventions — Oxaliplatin; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OXP (Experimental): Oxaliplatin 130mg/m2 + 5DW 500ml MIV over 2HR D1 Prednisolone 100mg/Day D1-D5 Every 3 weeks Maximum 6 cycles of treatment will be given for this study. Subjects will be treated for at least 1 cycle and to a maximum of 6 cycles unless there is documented disease progression, unacceptable adverse events or withdrawal of consent.
  Interventions: Drug: Oxaliplatin, Prednisolone

INTERVENTIONS:
Drug: Oxaliplatin, Prednisolone — OXALIPLATIN+PREDNISOLONE (OX-P)
  D1 Oxaliplatin 130mg/m2 + 5DW 500ml MIV over 2hr
  D1-5 Prednisolone 40-30-30 mg/day P.O
  every 3 weeks

SUMMARY:
The investigators are willing to investigate the efficacy and safety of oxaliplatin and prednisolone (Ox-P) combination in patients with previously treated MZL who have a few clinical trial data.

DETAILED DESCRIPTION:
Over its long survival duration, MZL often involves frequent relapses. Overall, more than 50% of MZL patients experience a relapse within 10 years. However, Relapsed or refractory MZL represent a therapeutic dilemma in every day clinical practice and no prospective studies on large series have been published so far. The rarity of these disorders and some difficulties in the differential diagnosis from other low-grade lymphoma subtypes are obstacles in conducting epidemiological surveys and in properly describing clinical features and outcomes.

Oxaliplatin, a platinum coordination complex with an oxalato-ligand as the leaving group and a 1,2-diaminocyclohexane carrier, possesses higher cytotoxic potency on molar basis than cisplatin and carboplatin and was reported to be active in patients with NHL as a single agent. In addition, the substitution of cisplatin by oxaliplatin in the DHAP regimen, another commonly used one in relapsed or refractory NHL, showed meaningful antitumor activity with favourable toxicity profile.

In the previous phase II study of oxaliplatin for treatment of patients with mucosa-associated lymphoid tissue lymphoma, a total of 16 patients with MALT lymphoma of various sites of origin (four of the ocular adnexa, five of the salivary glands, three of the stomach, two of the lung, and one of the colon and the breast) were administered oxaliplatin at a dose of 130 mg/m2 infused during 2 hours every 3 weeks. Fifteen patients responded to chemotherapy, with nine achieving CR (56%), six (37.5%) achieving partial response, and one achieving stable disease; the median time to response was 4 months (range; 2 to 4 months).

Based upon the promising results of oxaliplatin regimen in refractory NHL and first-line treatment of MZL, The investigators are willing to investigate the efficacy and safety of oxaliplatin and prednisolone (Ox-P) combination in patients with previously treated MZL who have a few clinical trial data.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed marginal zone B-cell lymphomas
* Failure to achieve a clinical benefit (≥SD) with the initial treatment, or recurrent disease
* Performance status (ECOG) ≤2
* Age ≥ 20
* At least one or more bi-dimensionally measurable lesion(s) defined as; ≥2 cm by conventional CT or ≥ 1 cm by spiral CT or skin lesion (photographs should be taken) or measurable lesion by physical examination
* Adequate kidney functions defined as; Cr < 2.0 mg% or Ccr > 60 ml/min
* Adequate liver functions defined as; Transaminases < 3 X upper normal values; Bilirubin < 2 mg%
* Adequate bone marrow functions defined as; ANC > 1500/㎕, platelet > 75000/㎕
* Ann Arbor stage III or IV
* Ann Arbor stage I or II, which is not adequate for RT or surgical approach (e.g. multiple lung lesions, multiple colon involvement, remote abdominal LN with stomach involvement)
* Written informed consent approved by Institutional review board or Ethic committee

Exclusion Criteria:

* Any other malignancies within the past 5 years except skin basal cell ca or CIS of cervix
* Serious co-morbid diseases
* Pregnancy or breast feeding
* Previous history of drug allergy to one of the drugs in the study regimen
* During this study duration, patients who take other clinical trial medication, chemotherapy, hormonal therapy, or immunotherapy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2009-10; Primary Completion 2013-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Response rate by International Working Group Response Criteria | 6 month after treatment

SECONDARY OUTCOMES:
progression free survival | 3 year after start
overall survival | 5 year after start

CONTACTS AND LOCATIONS:
Overall Officials: Cheolwon Suh, M.D., Ph.D., Principal Investigator — Asan Medical Center; Sung Yong Oh, M.D., Ph.D., Study Director — Dong-A University
Locations (1):
- Dong-A University Hospital, Busan, South Korea

REFERENCES:
- [Derived] Oh SY, Kim WS, Kim JS, Chae YS, Lee GW, Eom HS, Ryoo HM, Lee S, Kim SJ, Yoon DH, Won JH, Hong J, Park J, Lee SM, Hong JY, Park E, Kim HJ, Yang DH, Kim HJ, Suh C. A phase II study of oxaliplatin and prednisone for patients with relapsed or refractory marginal zone lymphoma: Consortium for Improving Survival of Lymphoma trial. Leuk Lymphoma. 2016;57(6):1406-12. doi: 10.3109/10428194.2015.1099650. Epub 2015 Nov 16. PMID 26413982